CLINICAL TRIAL: NCT05233475
Title: Get Going After concussIonN Lite (GAIN Lite): A Digital Intervention to Reduce Impairing Post-concussional Mild-to-moderate Symptoms in Adults
Brief Title: Get Going After concussIonN Lite
Acronym: GAIN Lite
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Hammel Neurorehabilitation Centre and University Research Clinic (Other); Health Research Foundation of Central Denmark Region (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100276
Record Dates: First submitted 2022-01-10; First posted 2022-02-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-05

CONDITIONS: Brain Concussion; Mild Traumatic Brain Injury; Commotio Cerebri
Keywords: Brain concussion; Behavior therapy; Early intervention; Mild traumatic brain injury; Post-concussion syndrome; Rivermead post-concussion symptoms questionaire
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome

STUDY DESIGN:
Intervention Model Description: Feasibility study, randomized controlled trial, implementation study and a prospective cohort study.
Who Masked: Care Provider
Masking Description: Both groups will recieve enhanced usual care. The care providers providing the enhanced usual care, will be blinded to group assignment. As the outcome assessor are the participants when the outcome is participant-reported outcomes, none of the outcome assessors are blinded, as it is impossible to blind the participants to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (EUC) (Active Comparator): Enhanced usual care (EUC):
  All participants will by a health professional be shortly informed about the typical recovery process, the given reassurance about the prognosis.as well as advice on adaptive illness behaviours post-concussion.
  Interventions: Behavioral: Enhanced usual care (EUC)
- Intervention Group (EUC + GAIN Lite) (Experimental): GAIN Lite:
  GAIN Lite in an add-on to EUC, and contains two major components: 1) self-administrated e-learning videos and 2) up to four hours video- or phone sessions with an allocated therapist (either an occupational- or a physiotherapist) during a period of 8 weeks. Health professionals provide feedback and guidance, addressing the specific aims and context of the individual.
  Interventions: Behavioral: Enhanced usual care (EUC); Behavioral: Get Going after concussIoN Lite

INTERVENTIONS:
Behavioral: Enhanced usual care (EUC) — Enhanced usual care (EUC):
  All participants will by a health professional be shortly informed about the typical recovery process, the given reassurance about the prognosis.as well as advice on adaptive illness behaviours post-concussion.
Behavioral: Get Going after concussIoN Lite — GAIN Lite:
  GAIN Lite in an add-on to EUC, and contains two major components: 1) self-administrated e-learning videos and 2) up to four hours video- or phone sessions with an allocated therapist (either an occupational- or a physiotherapist) during a period of 8 weeks. Health professionals provide feedback and guidance, addressing the specific aims and context of the individual.
  Other Names: GAIN Lite; KORT OG GODT OM HJERNERYSTELSE
  Arms: Intervention Group (EUC + GAIN Lite)

SUMMARY:
Background:

Concussion affects around 25 000 people each year in Denmark. A large research initiative (GAIN 2.0) has been established, and the current study is a part of this initiative.

Aims:

1. To develop and test the efficacy of a novel intervention for people with persistent post-concussional mild-to-moderate symptoms: "Get going After concussion Lite" (GAIN Lite).
2. To increase the knowledge about the target group by investigating the association of physical activity, digital behaviour, and symptom load.

Methods:

A randomized controlled trial, comparing GAIN Lite to enhanced usual care. 100 adults diagnosed with a concussion at hospitals in Central Denmark Region or referred from general practitioners will be recruited. GAIN Lite is a digital intervention, and the primary outcome is the severity of post-concussional symptoms. A prospective cohort study will be performed to investigate the association between physical activity, cognitive processing, and symptom load.

DETAILED DESCRIPTION:
Get going After concussIonN Lite (GAIN Lite): An digital intervention to reduce impairing post-concussional mild-to-moderate symptoms in adults

Background:

Concussion, the mildest form of traumatic brain injury, is an important public health concern, affecting around 25 000 people each year in Denmark. Symptoms are associated with high societal burden due to the long-term impact on labour market attachment and increased health care usage and social welfare benefits. Evidence for effective treatment strategies is scarce, resulting in only weak recommendations for most treatment approaches, as reflected in the recently published National Guidelines for Non-Pharmacological treatment for post-concussion symptoms (PCS). Recently, the effect of a novel intervention "Get going After concussIoN" (GAIN) for people with persistent severe PCS was examined with promising results. Based on GAIN, a large research initiative (GAIN 2.0), has been established, and the present study is a part of this initiative.

Aims

1. To develop and test the efficacy of a digital intervention for people with persistent mild-to-moderate PCS: "Get going After concussion Lite" (GAIN Lite).
2. To increase the knowledge about the target group by investigating the association of physical activity, digital behaviour, and symptom load.

Primary hypothesis:

Participants receiving GAIN Lite will 3 months after end of treatment report statistically and clinically significantly greater reduction of PCS compared to participants receiving enhanced usual care.

Methods:

The present study is a randomized controlled trial (RCT), comparing GAIN Lite to enhanced usual care. GAIN Lite is characterized as a complex intervention as described by the UK Medical Research Council (MRC) guidelines. Accordingly, GAIN Lite will be developed, feasibility-tested and evaluated before implementation into the RCT. Furthermore, the ADAPT process model outlined by Moore et al. will guide the process. During the RCT, a mixed-methods evaluation will be performed to evaluate the cost-effectiveness of GAIN Lite and to identify prerequisites for clinical implementation. Furthermore, a prospective cohort study will be performed to investigate which features of digital behaviour are related to symptom load and physical activity. The project is conducted in the Central Denmark Region and led by Hammel Neurorehabilitation Centre and University Research Clinic. One hundred people between the age of 18-60 diagnosed with a concussion at public hospitals in the Central Denmark Region will be identified from an administrative hospital register. In addition, participants can be referred to the study by general practitioners. Potential participants will approx. 2 months after the concussion receive a standardised and validated battery of questionnaires measuring PCS and daily functioning. Participants considered likely to meet the inclusion criteria will be invited to further screening for eligibility by a physician. Eligible participants will be randomised by a computer algorithm with predefined concealed random numbers to either 1) Enhanced usual care (EUC) or 2) GAIN Lite added to EUC. EUC consists of short information by a health professionel about the typical recovery process, the given reassurance about the prognosis as well as advice on adaptive illness behaviours post-concussion. GAIN Lite is a digital program that contains two major components: 1) self-administrated e-learning videos , and 2) up to four hours video- or phone sessions with an allocated therapist (either an occupational- or a physiotherapist) during a period of 8 weeks. The intervention begins 2-4 months after the onset of the concussion. The primary outcome is PCS measured by Rivermead Postconcussion Questionnaire (RPQ). All participants will complete self-reported measures at baseline, at end of treatment and 3 and 6 months after end of treatment. In a subgroup, an app will monitor digital behaviour on the participants' smartphones for 6 months. During the same period, participants will be frequently asked to rate their PCS. Physical activity will be assessed with thigh-worn accelerometers regarding step counts, sedentary behaviour, and sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Concussion caused by a head trauma according to the diagnostic criteria recommended by the Danish Consensus Report on Commotio Cerebri (26). The criteria are based on recommendations by the WHO Task Force, but with the amendment, that there must have been a direct contact between the head and an object in order to rule out acceleration - deceleration traumas;
2. Age 18 to 60 years at the time of the trauma;
3. A total score of 10-30 on RPQ within 1 week before enrolment in the study;
4. Able to understand, speak and read Danish;
5. Living in Central Denmark Region;
6. Identified from registers of the emergency departments or referred by GPs to GAIN Lite within 2-4 months after a concussion

Exclusion Criteria:

1. Objective neurological findings and/or acute trauma CT scan indicating neurological disease or brain damage linked to the concussion, if performed;
2. Previous concussion within the last 2 years with ongoing PCS at the time of the present concussion
3. Severe misuse of alcohol, prescription drugs and/or illegal drugs
4. Severe psychiatric co-morbidity (e.g. bipolar disorder, autism, psychotic disorder (life time)) or severe neurological disease (e.g. multiple sclerosis) that impedes participation in the programme.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Rivermead Post-concussion Questionnaire (RPQ/DK) | 6 months: From baseline to 24 weeks after baseline
  RPQ/DK is a self-report questionaire to measure the severity of post-concussion symptoms covering physical, cognitive, and emotional symptoms with 16 sub-items and a total sum score (range 0-64, higher score define more severe status)
Utrecht Scale for Evaluation of Rehabilitation-Participation (USER-P/DK) | 6 months: From baseline to 24 weeks after baseline
  USER-P/DK is a self-report questionaire that covers aspects of participation with three separate scales: Frequency, Restrictions and Satisfaction. The restrictions scale will be used. It contains 11 sub-items that are based on whether the participant experience any limitations in daily life. A sum score from 0-100 i created. (A higher score indicates a more favorable level of participation, i.e. fewer restrictions experienced.)

SECONDARY OUTCOMES:
Brief Illness Perception Questionnaire (B-IPQ/DK) | 3 months: From baseline to 12 weeks after baseline (End of treatment)
  B-IPQ/DK consists of nine self-reported items: Eight items that covers cognitive illness, emotional representations and illness comprehensibility on a 0-to-10 response scale. (Range 0-80, higher score reflects a more negative perception). Item 9 is an open-ended response item, which asks paticipants to list the three most important causal factors in their illness. Responses to the causal item can be grouped into categories and analysed.
Behavioral Response to Illness Questionnaire (BRIQ/DK) | 3 months: From baseline to 12 weeks after baseline (End of treatment)
  BRIQ/DK is a self-report measure to assess frequency of illness behaviors, and consists of 4 subscales (19 items) on a 0-5 response scale (Range 0-95, higher scores indicate that the participant engaged in the behavior more frequently)
Treatment Inventory of Costs in Patients with psychiatric disorders (TiC-P) | 9 months: From baseline to 36 weeks after baseline
  TiC-P/DK is a self-report measure designed to assess direct and indirect costs associated with mental health. Part II collects information on respondents' workplace absenteeism and/ or reduction in productivity in paid or unpaid work due to mental health illnesses in the past month.
Work Ability Index Short form (WAI-2) | 9 months: From baseline to 36 weeks after baseline
  The WAI/DK describes how capable an employee is of doing his/her job and the questionnaire consists of seven subscales referring to these aspects of work ability: Subscale 1 is used (WAI 1: current work ability compared with lifetime best)

OTHER OUTCOMES:
Number of participants who receive no public assistance benefits (State education fund grants excepted) | Six months after end of treatment
  Register based data on employment in the Danish Register for Evaluation of Marginalisation (DREAM). This register contains weekly information on social transfer payments for all residents of Denmark (since 1996).
Number of participants who receive public assistance benefits related to illness in more than three consecutive weeks | Six months after end of treatment
  Register based data on long term sick leave in the Danish Register for Evaluation of Marginalisation (DREAM). This register contains weekly information on social transfer payments for all residents of Denmark (since 1996).
The degree of employment (based on whether labor market contributions have been paid) | Six months after end of treatment
  Register based data job stability in the Danish Register for Evaluation of Marginalisation (DREAM). This register contains weekly information on social transfer payments for all residents of Denmark (since 1996).
Continuously recording the interaction of 50 participants with their smartphones during a period of 3 months (The smart phone use will be linked to activity level and PCS) | Three months
  Touchscreen data will be gathered in the background with an app (TapCounter) installed on the participants smart phones (Android users only due to system restrictions). The off-the-shelf data gathering tool available through QuantActions, Lausanne will be used. Raw smartphone taps will be converted into candidate measures for health, such as (i) Tapping speed; (ii) Typing speed; (iii) The speed of entering a passcode; (iv) The speed of finding an App icon on the home screen; (v) The number of interactions
Continuously collecting seven days of accelerometer-assessed physical activity in 50 participants once a month for three months (The activity level will be linked to PCS and smart phone use) | Once a month for three months
  Physical activity will be assessed with thigh-worn accelerometers (Axivity, Ltd, Newcastle AX3) regarding step counts, sedentary behaviour, and sleep
Post-concussion symptoms (PCS) is measures on the Rivermead Post-concussion Questionnaire (RPQ/DK) in 50 participants once a month for three months (PCS will be linked to smart phone use and activity level) | Once a month for three months
  RPQ/DK is a self-report questionaire to measure the severity of PCS covering physical, cognitive, and emotional symptoms with 16 sub-items and a total sum score (range 0-64, higher score define more severe status)
Evaluation of the feasibility, acceptability, and tolerability of the intervention will be made during the feasibility phase. Individual, organizational, and structural aspects of clinical implementation will be evaluated at the end of the RCT | Before implemention into the RCT and before implementation into clinical practice
  Semi-structured interviews will be used to evaluate the experiences of all involved stakeholders (participants, professionals, developers, and management).

CONTACTS AND LOCATIONS:
Overall Officials: Sedsel Pedersen, PhD student, Principal Investigator — Hammel Neurorehabilitation Centre and University Research Clinic
Locations (1):
- Hammel Neurorehabilitation Centre and University Research Clinic, Hammel, Deb´nmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pedersen SKS, Thastum MM, Odgaard L, Naess-Schmidt ET, Pedersen CB, Nygaard C, Pallesen H, Silverberg ND, Brunner I. A remotely delivered intervention targeting adults with persisting mild-to-moderate post-concussion symptoms (GAIN Lite): a study protocol for a parallel group randomised trial. Trials. 2024 Oct 26;25(1):720. doi: 10.1186/s13063-024-08546-3. PMID 39456081
- [Background] Thastum MM, Rask CU, Naess-Schmidt ET, Tuborgh A, Jensen JS, Svendsen SW, Nielsen JF, Schroder A. Novel interdisciplinary intervention, GAIN, vs. enhanced usual care to reduce high levels of post-concussion symptoms in adolescents and young adults 2-6 months post-injury: A randomised trial. EClinicalMedicine. 2019 Dec 16;17:100214. doi: 10.1016/j.eclinm.2019.11.007. eCollection 2019 Dec. PMID 31891145
- [Background] Naess-Schmidt ET, Thastum MM, Stabel HH, Odgaard L, Pedersen AR, Rask CU, Silverberg ND, Schroder A, Nielsen JF. Interdisciplinary intervention (GAIN) for adults with post-concussion symptoms: a study protocol for a stepped-wedge cluster randomised trial. Trials. 2022 Jul 29;23(1):613. doi: 10.1186/s13063-022-06572-7. PMID 35906645